CLINICAL TRIAL: NCT03470662
Title: Effect of Prospective Care Bundle on Prevention of Delirium Among Elderly Patients With Hip Fractures
Brief Title: Prevention of Delirium Among Elderly Patients With Hip Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhoupu Hospital, Pudong New Area, Shanghai, China (Other)
Responsible Party: Principal Investigator, Xiaoxiao Zhou, Director of Orthopaedics Department, Zhoupu Hospital, Pudong New Area, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YuFengbinDelirium
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Delirium; Hip Fractures
Keywords: Hip fractures; Delirium; Aged; Care bundle
MeSH Terms: conditions — Delirium; Hip Fractures | interventions — Patient Care Bundles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Care bundle
  Interventions: Other: Care bundle
- control group (No Intervention): routine care

INTERVENTIONS:
Other: Care bundle — Care bundle
  Arms: experimental group

SUMMARY:
Objective: To evaluate the effect of care bundle on prevention of delirium among elderly patients with hip fractures.

Methods: A prospective randomized case control study was performed for 80 patients (≥65 years) with hip fractures treated surgically according to their ages and the type of fractures from March 1th of 2017 to June 30th of 2017．There were 11 males and 69 females, with the age of (79.3±7.84) years. Confusion assessment method (CAM) was applied to diagnose delirium after surgery, the subjects were randomized divided into experimental group (n=43) and control group (n=37). The parameters next were recorded and analyzed, including age, gender, type of fractures, type of internal instrument, amount of bleeding, time between injured to surgery, time length of operation, type of operation, VAS, incidence of delirium, perioperative complications and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years
* with hip fractures
* treated surgically

Exclusion Criteria:

* <65 years
* psychiatric history
* ICU post-operation
* refuse to join this study
* have delirium pre-operation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
incidence of delirium among elderly patients with hip fractures | 3 weeks
  study hypothesis: the incidence of delirium postoperatively in experimental group is lower compared with control group

CONTACTS AND LOCATIONS:
Locations (1):
- Zhoupu Hospital Shanghai, Shanghai, China